CLINICAL TRIAL: NCT02311998
Title: A Phase I/II Study of Bosutinib in Combination With Inotuzumab Ozogamicin in CD22-Positive Philadelphia-Chromosome Positive Acute Lymphoblastic Leukemia and Chronic Myeloid Leukemia Lymphoid Blast Phase
Brief Title: Phase I/II Study of Bosutinib in Combination With Inotuzumab Ozogamicin in CD22-positive PC Positive ALL and CML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0435; NCI-2014-02606 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0435 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Blasts More Than 5 Percent of Bone Marrow Nucleated Cells; CD22 Positive; Philadelphia Chromosome Positive, BCR-ABL1 Positive Chronic Myelogenous Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive
MeSH Terms: conditions — Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib; Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment (bosutinib, inotuzumab ozogamicin) Phase I Dose 1 (Experimental): Patients receive bosutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Patients with confirmed CR, CRi, CCyR and/or absence of MRD may receive inotuzumab ozogamicin IV on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosutinib; Biological: Inotuzumab Ozogamicin
- Treatment (bosutinib, inotuzumab ozogamicin) Phase II (Experimental): Patients receive bosutinib at the Maximum Tolerated Dose from the Phase I dose part, PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Patients with confirmed CR, CRi, CCyR and/or absence of MRD may receive inotuzumab ozogamicin IV on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosutinib; Biological: Inotuzumab Ozogamicin
- Treatment (bosutinib, inotuzumab ozogamicin) Phase I Dose 2 (Experimental): Patients receive bosutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Patients with confirmed CR, CRi, CCyR and/or absence of MRD may receive inotuzumab ozogamicin IV on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosutinib; Biological: Inotuzumab Ozogamicin
- Treatment (bosutinib, inotuzumab ozogamicin) Phase I Dose 3 (Experimental): Patients receive bosutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Patients with confirmed CR, CRi, CCyR and/or absence of MRD may receive inotuzumab ozogamicin IV on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosutinib; Biological: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Bosutinib — Given PO
  Other Names: Bosulif; SKI 606; SKI-606
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC-544; Way 207294; WAY-207294

SUMMARY:
This phase I/II trial studies the side effects and best dose of bosutinib when given together with inotuzumab ozogamicin and to see how well it works in treating patients with acute lymphoblastic leukemia or chronic myeloid leukemia that has come back or does not respond to treatment. Bosutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotoxins, such as inotuzumab ozogamicin, are antibodies linked to a toxic substance and may help find cancer cells that express CD22 and kill them without harming normal cells. Giving bosutinib together with inotuzumab ozogamicin may be a better treatment for acute lymphoblastic leukemia or chronic myeloid leukemia.

DETAILED DESCRIPTION:
If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study and whether or not you have received earlier treatment for leukemia. Up to 36 participants will be enrolled in Part 1 of the study, and up to 44 participants will be enrolled in Part 2.

If you are enrolled in Part 2, you will receive bosutinib at the highest dose that was tolerated in Part 1. All participants in Parts 1 and 2 will receive the same dose of inotuzumab ozogamicin.

Study Drug Administration. You will take bosutinib tablets by mouth 1 time each day with food. If you miss or vomit a dose of bosutinib, do not take "make up" the dose. Wait and take your next dose as scheduled the next day.

You will also receive inotuzumab ozogamicin by vein over about 1 hour on Days 1, 8, and 15 of each 28-day cycle. If the doctor thinks it is needed, you may switch to a different dosing schedule and receive inotuzumab ozogamicin 1 time every 4 weeks.

You will be given standard drugs (such as acetaminophen/paracetamol, antihistamines, and/or steroids) to help decrease the risk of side effects. If your doctor thinks it is needed, you may also receive hydroxyurea to control your white blood cell count while you are on study. You may ask the study staff for information about how these drugs are given and their risks.

Follow-Up After your end-of-treatment visit or call, you will be called 1 time about every 12 weeks (for up to 1 year) and asked about any anti-cancer therapy you may have started. This call will last about 5 minutes.

After completion of study treatment, patients are followed up every 12 weeks for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory B-cell ALL or CML in lymphoid blast phase; Philadelphia chromosome must be present at screening (as determined by cytogenetic analysis, fluorescence in situ hybridization [FISH], or polymerase chain reaction [PCR] [i.e., BCR-ABL positive]); Note: patients with CML who have received treatment with tyrosine kinase inhibitors for their CML, and have progressed to lymphoid blast phase are eligible for frontline treatment; Frontline Ph+ ALL or CML-lymphoid blast phase (LBC) Cohort: Patients with newly-diagnosed Ph+ ALL or CML-LBC, who have received no or minimal treatment (minimal treatment is defined as treatment with steroids/hydroxyurea of =< 2 week duration; vincristine =< 2 doses; tyrosine kinase inhibitor of =< 4 week duration; =< 2 doses of cytarabine) and are >= 60 years or older are eligible; patients must have bone marrow blasts > 5% at the time of screening
* Expression of CD-22 in >= 20% blasts
* Eastern Cooperative Oncology Group (ECOG) performance status score of < or = 2
* Serum bilirubin < or = 2.0 mg/dl
* Serum creatinine < or = 2.0 mg/dl
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < or = 3 x upper limit of normal (ULN)
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (beta-hCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 30 days following the last dose of study drug; effective methods of birth control include: birth control pills, shots, implants (placed under the skin by a health care provider) or patches (placed on the skin); intrauterine devices (IUDs); condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide; females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years; patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses)
* Patients with active unstable angina, concomitant clinically significant active arrhythmias, myocardial infarction within 6 months, or congestive heart failure New York Heart Association class III-IV; patients with a cardiac ejection fraction (as measured by either multi gated acquisition scan [MUGA] or echocardiogram) < 40% are excluded
* Known evidence of active cerebral/meningeal disease; patients may have history of central nervous system (CNS) leukemic involvement if definitively treated with prior therapy and no evidence of active disease (defined as >= 2 consecutive spinal fluid assessments with no evidence of disease) at that time of registration
* Previous treatment with any anti-CD22 directed therapy
* Patients with previous allogeneic stem cell transplant (SCT) if they meet either of the following criteria:

  * < 100 days from allogeneic SCT
  * Active acute or chronic graft-versus-host disease (GvHD), or
  * Receiving immunosuppressive therapy as treatment for GvHD within the last 7 days
* Patients with uncontrolled active infections (viral, bacterial, or fungal) are not eligible
* Active hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Patients with liver cirrhosis or other serious active liver disease or with suspected alcohol abuse
* History of autoimmune diseases (such as systemic lupus erythematosus [SLE], Wegener's, Wegener's granulomatosis, polyarteritis nodosa); Note: Prior autoimmune diseases are allowed as long as clinically stable
* Prior chemotherapy/radiotherapy/investigational therapy within 2 weeks before the start of study drugs with the following exceptions:

  * To reduce the circulating lymphoblast count or palliation: steroids, hydroxyurea; no washout necessary for these agents
  * For ALL maintenance/CML treatment: mercaptopurine, methotrexate, vincristine, single-agent, single-dose of cytarabine and/or tyrosine kinase inhibitors; these agents should be discontinued at least 48 hours prior to start of study drugs; (Note: the interval of time from last dose of any approved tyrosine kinase inhibitor [TKI] to start of protocol treatment is 48 hours regardless of the indication for treatment with the TKI)
* Patients who have not recovered from acute non hematologic toxicity (to =< grade 1) of all previous therapy prior to enrollment
* Females who are pregnant or lactating
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study
* Patients previously exposed to bosutinib are eligible unless they carry T315I
* Patients with T315I mutations will be excluded (this criteria is not applicable for the frontline Ph+ ALL or CML-LBC cohort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1: Patients receive bosutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Patients with confirmed CR, CRi, CCyR and/or absence of MRD may receive inotuzumab ozogamicin IV on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Bosutinib: Given PO 300mg
  Inotuzumab Ozogamicin: Given IV
- Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2: Patients receive bosutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Patients with confirmed CR, CRi, CCyR and/or absence of MRD may receive inotuzumab ozogamicin IV on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Bosutinib: Given PO 400mg
  Inotuzumab Ozogamicin: Given IV
- Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3: Patients receive bosutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Patients with confirmed CR, CRi, CCyR and/or absence of MRD may receive inotuzumab ozogamicin IV on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Bosutinib: Given PO 500mg
  Inotuzumab Ozogamicin: Given IV
Period: Overall Study
Arm/Group | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase II
Started | 3 | 6 | 9 | 4
Completed | 3 | 6 | 9 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase II | Total
Number analyzed (Participants) | 3 | 6 | 9 | 4 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 7 | 1 | 14
  >=65 years | 1 | 2 | 2 | 3 | 8
Age, Continuous [Median (Full Range); unit: years] | 43 [27 to 66] | 60 [35 to 74] | 63 [19 to 69] | 71 [62 to 81] | 64 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 2 | 12
  Male | 1 | 3 | 4 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 6 | 9 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Bosutinib All Phase I Participants
Description: Maximum tolerated dose of bosutinib defined as the highest dose level in which < 2 patients of 6 develop first course dose limiting toxicity (Phase I). Dose levels assessed were dose 1 = 300 mg, dose 2 = 400 mg, and dose 3 = 500 mg.
Time Frame: At day 28
Population: This outcome is only intended for the Phase I arm of this study
Measure: Number; unit: Milligrams
Arm/Group | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1
Number analyzed (Participants) | 18
Milligrams | 400

2. Primary Outcome: Number of Participants With a Major Hematologic Response
Description: Major Hematologic Response i(MaHR) is defined as Complete Response (CR) + Complete Remission without Incomplete Blood Count Recovery (CRi). CR was defined as absence of circulating blasts with bone marrow blasts <5% and recovery of neutrophil count to ≥1.0 x 10^9/L and platelet count to ≥100 x10^9/L. The CRi was defined as meeting criteria for CR except for neutrophil and/or platelet recovery. Response was assessed by bone marrow analysis after each cycle of therapy until attainment of CR/CRi.
Time Frame: Up to 6 years, 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase II
Number analyzed (Participants) | 3 | 6 | 9 | 4
Participants | 3 | 4 | 8 | 4

3. Secondary Outcome: Duration of Response
Description: Estimated using the method of Kaplan-Meier. Response date to loss of response or last follow up.
Time Frame: Up to 6 years, 11 months
Population: Of the 18 participants treated during Phase I, 15 were evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase II
Number analyzed (Participants) | 3 | 6 | 9 | 4
Months | 4.1 [1.9 to 8.8] | 7.7 [6.2 to 73.8] | 27.2 [2.1 to 68.9] | 5.1 [0.7 to 8.1]

4. Secondary Outcome: Overall Survival (OS)
Description: Estimated using the method of Kaplan-Meier. Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 6 years, 11 months
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase II
Number analyzed (Participants) | 3 | 6 | 9 | 4
Months | 8.2 [6.8 to 10.7] | 9.6 [2.0 to 74.6] | 47.5 [2.7 to 72.8] | 5.3 [2.0 to 28.2]

ADVERSE EVENTS:
Time Frame: Up to 6 years, 11 months.
Arm/Group | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3 | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase II
All-Cause Mortality (participants affected / at risk) | 3/3 | 5/6 | 4/9 | 2/4
Serious Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 5/9 | 4/4
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 8/9 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1 (N=3) | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2 (N=6) | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3 (N=9) | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase II (N=4)
Abdominal pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 1 (N=3) | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 2 (N=6) | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase I Dose 3 (N=9) | Treatment (Bosutinib, Inotuzumab Ozogamicin) Phase II (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain cardiac (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blisters Lip (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Eye disorders (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Deconditioning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Flushing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (General disorders) | 2 (2) | 1 (3) | 1 (1) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
hepatosplenomegaly (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 4 (4) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0) | 0 | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
mild lip swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4) | 3 (3)
Nervous system disorders (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
night sweats (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Rash maculo papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 2 (3) | 4 (4) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02311998/Prot_SAP_000.pdf